CLINICAL TRIAL: NCT01967914
Title: Can Plethysmography Variability Index (PVI) Predict Spinal Induced Hypotension in Women Undergoing Cesarean Delivery?
Brief Title: PVI for Prediction of Spinal Induced Hypotension
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00046443
Record Dates: First submitted 2013-10-17; First posted 2013-10-23 (Estimated); Last update posted 2015-06-17 (Estimated); Status verified 2015-06

CONDITIONS: Spinal Induced Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Women undergoing cesarean delivery under spinal anesthesia
  Interventions: Other: PVI

INTERVENTIONS:
Other: PVI — Measurement of PVI (plethysmography variability index)

SUMMARY:
The hypothesis is that plethysmography variability index can predict the occurrence of hypotension after spinal anesthesia for cesarean delivery

ELIGIBILITY:
Inclusion Criteria:

* English speaking ASA I-II non-laboring women with single gestations ≥36 weeks
* Scheduled or unscheduled cesarean delivery under spinal anesthesia
* Height: 5 feet-5 feet 11 in.

Exclusion Criteria:

* Laboring women needing an emergency cesarean delivery
* Severe hypertensive disease of pregnancy defined as systolic blood pressure (SBP)>160mmHg, diastolic blood pressure (DBP)>110mmHg requiring antihypertensive treatment or associated with significant proteinuria.
* Severe Cardiac disease in pregnancy with marked functional limitations
* Diabetes type I
* Patients on Monoamine Oxidase Inhibitors or Tricyclic Antidepressants
* Inclusion in another anesthetic study involving drug administration.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women undergoing cesarean delivery under spinal anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2013-10; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Correlation between baseline PVI and change in SBP from baseline. | Intraoperative (approximately 2 hours)
  Correlation between baseline PVI and change in SBP from baseline.

SECONDARY OUTCOMES:
Correlation between plethysmography variability index (PVI) change in response to passive leg raising (PLR) and change in SBP and pulse rate (PR) from baseline, and need for vasopressors | Intraoperative (approximately 2 hours)
  Correlation between PVI change in response to PLR and change in SBP and pulse rate (PR) from baseline, and need for vasopressors
Correlation between intraoperative PVI change from baseline with change in SBP and PR from baseline, and need for vasopressors. | Intraoperative (approximately 2 hours)
Correlation between baseline PVI and need for vasopressors. | Intraoperative (approximately 2 hours)
Correlation between baseline PVI and change in SBP and PR from baseline. | Intraoperative (approximately 2 hours)
Correlation between CO change in response to SLR with change in SBP and PR from baseline, and need for vasopressors | Intraoperative (approximately 2 hours)

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf S Habib, MB, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States